CLINICAL TRIAL: NCT05886907
Title: Assessing the Clinical Performance of Two Frequent Replacement Silicone Hydrogel Multifocal Toric Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLR624-M103
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Refractive Errors; Presbyopia; Astigmatism
Keywords: Contact Lenses
MeSH Terms: conditions — Refractive Errors; Presbyopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Subjects will wear the products (test and comparator) in a predetermined order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID223188, then Ultra MFT (Other): Lehfilcon A multifocal toric contact lenses worn first, with samfilcon A multifocal toric contact lenses worn second. Each product will be worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE will be used for daily contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal toric contact lenses; Device: Samfilcon A multifocal toric contact lenses; Device: CLEAR CARE
- Ultra MFT, then LID223188 (Other): Samfilcon A multifocal toric contact lenses worn first, with lehfilcon A multifocal toric contact lenses worn second. Each product will be worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE will be used for daily contact lens cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal toric contact lenses; Device: Samfilcon A multifocal toric contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A multifocal toric contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: LID223188
Device: Samfilcon A multifocal toric contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: Ultra MFT; Bausch + Lomb Ultra® Multifocal for Astigmatism
Device: CLEAR CARE — Hydrogen peroxide based contact lens cleaning and disinfecting solution
  Other Names: CLEAR CARE® Cleaning and Disinfecting Solution

SUMMARY:
The purpose of this clinical trial is to assess on-eye performance and overall fit of an investigational multifocal toric contact lens to aid in confirmation of the study lens design.

DETAILED DESCRIPTION:
Subjects will attend 3 study visits with a planned individual duration of participation of up to 10 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Requires ADD (additional power for near vision);
* Currently wears multifocal soft contact lenses in both eyes during the past 3 months;
* Manifest cylinder power between -0.75 diopter (D) and -1.00 D;
* Best Corrected Visual Acuity (BCVA) of logMAR 0.10 (Snellen 20/25) or better in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Current or history of pathologically dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear;
* Monovision contact lens wear.
* Other protocol-specified exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, CRD Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Johns Creek Research Clinic, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 investigative site located in the United States.
Pre-assignment Details: Of the 18 enrolled, 9 were exited prior to study lens assignment as screen failures. This reporting group includes all participants exposed to any study lenses evaluated in this study (9).
Groups:
- LID223188, Then Ultra MFT: Lehfilcon A multifocal toric contact lenses worn first, with samfilcon A multifocal toric contact lenses worn second. Each product was worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
- Ultra MFT, Then LID223188: Samfilcon A multifocal toric contact lenses worn first, with lehfilcon A multifocal toric contact lenses worn second. Each product was worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
Period: First Wear Period (Approx. 2 Days)
Arm/Group | LID223188, Then Ultra MFT | Ultra MFT, Then LID223188
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Wear Period (Approx. 2 Days)
Arm/Group | LID223188, Then Ultra MFT | Ultra MFT, Then LID223188
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID223188, Then Ultra MFT | Ultra MFT, Then LID223188 | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.0) | 65.0 (3.2) | 61.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1 | 4 | 5
  Black or African American | 3 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Visual Acuity (VA) With Study Lenses
Description: Visual Acuity (VA) was assessed binocularly (both eyes together) with study lenses in place at a distance of 4 meters using letter charts. VA was recorded in logarithm minimum angle of resolution (logMAR), where 0.0 logMAR equates to 20/20 Snellen (normal distance eyesight). A lower number indicates better visual acuity. No hypothesis testing is pre-specified for this endpoint.
Time Frame: Day 2, each wear period. A wear period was approximately 2 days.
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- LID223188: Lehfilcon A multifocal toric contact lenses worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
- Ultra MFT: Samfilcon A multifocal toric contact lenses worn bilaterally (in both eyes) during waking hours for approximately 2 days. CLEAR CARE was used for daily contact lens cleaning and disinfection.
Arm/Group | LID223188 | Ultra MFT
Number analyzed (Participants) | 9 | 9
logMAR | -0.04 (0.09) | -0.09 (0.07)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to 10 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study. The Other (Not Including Serious) Adverse Event table reports only the AEs that occurred above a 5% threshold in one or more arms.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID223188 Ocular; LID223188 Nonocular: Events reported in this group occurred while exposed to lehfilcon A multifocal toric contact lenses.
- Ultra MFT Ocular; Ultra MFT Nonocular: Events reported in this group occurred while exposed to samfilcon A multifocal toric contact lenses.
Arm/Group | Pretreatment | LID223188 Ocular | LID223188 Nonocular | Ultra MFT Ocular | Ultra MFT Nonocular
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/18 | 0/9 | 0/18 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/18 | 0/9 | 0/18 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/18 | 0/9 | 0/18 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT05886907/Prot_SAP_000.pdf